CLINICAL TRIAL: NCT00300950
Title: A Phase 2 Double-Blind, Placebo Controlled, Multi-center Adjuvant Trial of the Efficacy, Immunogenicity, and Safety of GI-4000; an Inactivated Recombinant Saccharomyces Cerevisiae Expressing Mutant Ras Protein Combined With a Gemcitabine Regimen Versus a Gemcitabine Regimen With Placebo, in Patients With Post-resection R0/R1 Pancreatic Cancer With Tumor Sequence Confirmation of Ras Mutations.
Brief Title: Safety and Efficacy of the Therapeutic Vaccine GI-4000 in Combination With Gemcitabine Versus Placebo for the Treatment of Non-metastatic, Post-resection Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlobeImmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: GI-4000-02
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Pancreas Cancer
Keywords: Pancreas Cancer; resected pancreas cancer; non-metastatic pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Gencitabine
  Interventions: Biological: GI-4000
- 2 (Experimental): Gemcitabine with GI-4000
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Biological: GI-4000 — Heat-killed yeast cell transfected with target ras mutation.
  Arms: 1
Drug: Gemcitabine — Chemotherapy
  Arms: 2

SUMMARY:
The GI-4000 therapeutic vaccine or placebo will be injected under the skin of post-resection, non-metastatic pancreas cancer patients. Patients will be monitored for recurrence as well as safety, and immune responses related to the injections.

ELIGIBILITY:
(A few general items required)

Inclusion Criteria:

* Patients with non-metastatic pancreas cancer post-resection that have a product-related ras mutation
* >18 years of age
* Negative skin test for hypersensitivity to Saccharomyces cerevisiae

Exclusion Criteria:

* Metastatic pancreas cancer patients post-resection
* Patients with no product-related ras mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2006-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Recurrence free time and survival | 5 years

CONTACTS AND LOCATIONS:
Locations (28):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tower Cancer Research Foundation, Beverly Hills, California
  - University of California San Diego, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Georgetown University Medical Center / Lombardi Cancer Center, Washington D.C., District of Columbia
  - Rush University Medical School, Chicago, Illinois
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - State University of NY at Stony Brook, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Texas Oncology, PA, Dallas, Texas
  - The Texas Cancer Center Dallas Southwest, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Froedtert Multi-Disciplinary Cancer Clinic, Milwaukee, Wisconsin
- India (10):
  - PSG Hospitals, Peelamedu, Coimbatore, Tamil Nadu
  - Sri Ramchandra Medical College & Research Institute, Ponur, Chennai, Tamil Nadu
  - Indo American Cancer Hospital and Research Centre, Hyderabad
  - KMC Hospital, Mangalore
  - Govt Medical Colleg & Hospital, Nagpur
  - Lake Shore Hospital & Research Centre, Nettoor, Cochin
  - G B Pan Hospital & Maulana Azad Medical College, New Delhi
  - Nizam's Institute of Medical Sciences, Panjagutta, Hyderaba
  - Lifeline Multispecialty Hospital, Perungudi, Chennai
  - Regional Cancer Centre, Trivandrum

REFERENCES:
- [Derived] Muscarella P, Bekaii-Saab T, McIntyre K, Rosemurgy A, Ross SB, Richards DA, Fisher WE, Flynn PJ, Mattson A, Coeshott C, Roder H, Roder J, Harrell FE, Cohn A, Rodell TC, Apelian D. A Phase 2 Randomized Placebo-Controlled Adjuvant Trial of GI-4000, a Recombinant Yeast Expressing Mutated RAS Proteins in Patients with Resected Pancreas Cancer. J Pancreat Cancer. 2021 Mar 23;7(1):8-19. doi: 10.1089/pancan.2020.0021. eCollection 2021. PMID 33786412